CLINICAL TRIAL: NCT03798418
Title: Sarcopenia and Risk of Falls in Patients With Major Chronic Diseases - Effects of Therapeutic Exercise and Nutrition Intervention
Brief Title: Sarcopenia and Risk of Falls in Patients With Major Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCH-170208
Record Dates: First submitted 2018-12-28; First posted 2019-01-10 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Osteoporosis; Chronic Kidney Diseases; Cancer
Keywords: Sarcopenia; stroke; osteoporosis; chronic kidney disease; cancer; balance and gait; fall
MeSH Terms: conditions — Stroke; Osteoporosis; Renal Insufficiency, Chronic; Neoplasms; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Active Comparator): elastic band strengthening exercise
  Interventions: Behavioral: elastic band strengthening exercise
- exercise combine diet counseling group (Experimental): elastic band strengthening exercise combined diet counseling.
  Interventions: Behavioral: elastic band strengthening exercise; Dietary Supplement: diet counseling

INTERVENTIONS:
Behavioral: elastic band strengthening exercise — 2-3days per week(150min per week)
  Other Names: thera-band strengthening exercise
Dietary Supplement: diet counseling — each patients in this group will receive4-5times diet counseling
  Other Names: nutrition counseling
  Arms: exercise combine diet counseling group

SUMMARY:
The objective of this study is to investigate the effects of therapeutic exercise and nutrition intervention for sarcopenia and risk of falls in patients with major chronic diseases. The outcomes will be analyzed regarding muscle strength, quality, and volume, etc., balance and gait, bone density, body composition, fall and quality of life after the intervention.

DETAILED DESCRIPTION:
The main common chronic diseases in the elderly such as stroke, osteoporosis, chronic kidney disease and cancer, have been regarded as the fall high-risk patients. These patients are considered to be at risk for sarcopenia due to decreased exercise, nutritional status, and other reasons. Sarcopenia can be diagnosed and intervened effectively to delay the vicious cycle of health. Past studies have pointed out that in addition to drug intervention, treatment for sarcopenia must be accompanied by appropriate exercise and nutritional intervention (such as protein supplements, vitamin D) in order to achieve the best prevention and treatment.

ELIGIBILITY:
* Inclusion Criteria:

  1. 55-85 years old
  2. 3-6 months after onset
  3. walk independently for at least 10m
* Exclusion Criteria:

  1. lower limb Brunnstrom stage >5
  2. combine other neuropathy diseases
  3. significant deformity of lower limb include: Modified Ashworth scale(MAS) >3; contracture, fracture, chronic joint pain.
  4. joint arthroplasty
  5. unstable vital sign
  6. can not cooperate study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change of walking speed | baseline: before intervention; follow-up: 3 months after intervention
  distance: 6m, patients can walk with foor orthosis and assistive devices
Change of grip force | before intervention; follow-up: 3 months after intervention
  Use a grip force meter (kg) to test both hands for test 3 times
Change of postural sway displacement | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure the postural sway displacement (mm)
Change of postural sway velocity | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure the postural sway velocity (mm/s)
Change of postural sway area | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure the postural sway area (mm^2)
Change of step time | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: step time (ms)
Change of stance time | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: stance time (ms)
Change of swing time | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: swing time (ms)
Change of single support time | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: single support time (ms)
Change of double support time | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: double support time (ms)
Change of step length | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: step distance (mm)
Change of stance length | before intervention; follow-up: 3 months after intervention
  Use computerized dynography to measure spatial gait parameter: stance distance (mm)
Change of muscle thickness | before intervention; follow-up: 3 months after intervention
  Use ultrasound to assess muscles morphological parameter: thickness (mm). Target muscles include quadriceps, hamstring, anterior tibialis, gastrocnemius.
Change of muscle fiber length | before intervention; follow-up: 3 months after intervention
  Use ultrasound to assess muscles morphological parameter: fiber length (mm). Target muscles include quadriceps, hamstring, anterior tibialis, gastrocnemius.
Change of muscle fiber orientation angle | before intervention; follow-up: 3 months after intervention
  Use ultrasound to assess muscles morphological parameter: fiber orientation angle (degrees). Target muscles include quadriceps, hamstring, anterior tibialis, gastrocnemius.
Change of muscle cross section area | before intervention; follow-up: 3 months after intervention
  Use ultrasound to assess muscles morphological parameter: cross-sectional area (mm^2).
  Target muscles include quadriceps, hamstring, anterior tibialis, gastrocnemius.
Change of physiological cost index (PCI) | before intervention; follow-up: 3 months after intervention
  Heart rate (HR: beats/min) and walking speed (m/s) have been previously shown to be linearly related to oxygen uptake at sub-maximal exercise levels. Combination of these two parameters yields a single value in beats per meter, the physiological cost index (PCI). This is calculated as Working HR - Resting HR (beats/min) / Walking speed (m/s)
Change of international Quality of Life Assessment Short Form -36 (SF-36) | before intervention; follow-up: 3 months after intervention
  including 8 health concepts: (1) physical functioning, (2) role limitations because of physical health problems; (3) bodily pain, (4) social functioning, (5) general mental health (psychological distress and psychological wellbeing), (6) role limitations because of emotional problems, (7) vitality (energy/fatigue), (8) general health perceptions.
  Scoring: answers to each question are scored which are then summed and transformed to a 0 - 100 scale.
  The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change of amplitude of Muscle activity | before intervention; follow-up: 3 months after intervention
  use electromyography to measure the muscles activity in microvolts (uv) included quadriceps, hamstrings, tibialis anterior, gastrocnemius during subject walking in self-selected speed in 6 meters.

SECONDARY OUTCOMES:
Change of concentration of CRP (C-Reactive Protein) | before intervention; follow-up: 3 months after intervention
  The concentration of CRP in the blood test. CRP is used mainly as a marker of inflammation.
Change of concentration of ALB (Serum albumin) | before intervention; follow-up: 3 months after intervention
  The concentration of ALB in the blood test. Albumin is the most important contributor to the maintenance of plasma colloid oncotic pressure; deficiency results in edema.
Change of concentration of Glomerular Filtration Rate (GFR) | before intervention; follow-up: 3 months after intervention
  The concentration of GFR in the blood test. The glomerular filtration rate is the best test to measure the patient's level of kidney function and determine the stage of kidney disease. It can calculate it from the results of the blood creatinine test.
Change of concentration of Hemoglobin (Hb) | Time Frame: before intervention; follow-up: 3 months after intervention
  The concentration of Hb in the blood test.
Change of concentration of Glucose SPOT | Time Frame: before intervention; follow-up: 3 months after intervention
  The concentration of Glucose SPOT in the blood test. TheSpot glucose measurement in epidermal interstitial fluid appears to be a promising alternative to capillary blood glucose estimation
Change of concentration of Cholesterol | before intervention; follow-up: 3 months after intervention
  The concentration of Cholesterol in the blood test.
Change of concentration of Triglyceride | before intervention; follow-up: 3 months after intervention
  The concentration of Triglyceride in the blood test.
Change of concentration of Transferrin | before intervention; follow-up: 3 months after intervention
  The concentration of Transferrin in the blood test.
Change of Berg balance test (BBS) | before intervention; follow-up: 3 months after intervention
  including 14 items which are scored on a 5 points scale (0-4). The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.
  The item scores are summed, minimum score =0, maximum score = 56
Change of Fugl-Meyer Assessment (FMA) | before intervention; follow-up: 3 months after intervention
  Items are scored on a 3-point ordinal scale (0 = cannot perform; 1 = performs partially; 2 = performs fully) Maximum Score = 226 points The 5 domains assessed include, Motor function (UE maximum score = 66; LE maximum score = 34), Sensory function (maximum score = 24), Balance (maximum score = 14), Joint range of motion (maximum score = 44), Joint pain (maximum score = 44)
Change of Body Mass Index (BMI) | before intervention; follow-up: 3 months after intervention
  (body weight) kg/(height) m*(height)m
Change of Mini-mental state examination (MMSE) | before intervention; follow-up: 3 months after intervention
  It is an 11-question measure that tests five areas of cognitive function:
  orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
Change of Modified Ashworth scale (MAS) | before intervention; follow-up: 3 months after intervention
  measures resistance during passive soft-tissue stretching, the score is ranged from 0-4 0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Change of Muscle tone | before intervention; follow-up: 3 months after intervention
  measure the muscle tone (kg/m) under muscle resting. Target muscles are quadricep, hamstring, anterior tibialis, gastrocnemius.

CONTACTS AND LOCATIONS:
Overall Officials: Tasen Wei, Doctor, Study Director — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No
only for research

REFERENCES:
- [Background] Biolo G, Cederholm T, Muscaritoli M. Muscle contractile and metabolic dysfunction is a common feature of sarcopenia of aging and chronic diseases: from sarcopenic obesity to cachexia. Clin Nutr. 2014 Oct;33(5):737-48. doi: 10.1016/j.clnu.2014.03.007. Epub 2014 Mar 29. PMID 24785098
- [Background] Stapleton T, Ashburn A, Stack E. A pilot study of attention deficits, balance control and falls in the subacute stage following stroke. Clin Rehabil. 2001 Aug;15(4):437-44. doi: 10.1191/026921501678310243. PMID 11518445
- [Background] Hyndman D, Ashburn A, Stack E. Fall events among people with stroke living in the community: circumstances of falls and characteristics of fallers. Arch Phys Med Rehabil. 2002 Feb;83(2):165-70. doi: 10.1053/apmr.2002.28030. PMID 11833018
- [Background] Kutner NG, Zhang R, Huang Y, Wasse H. Falls among hemodialysis patients: potential opportunities for prevention? Clin Kidney J. 2014 Jun;7(3):257-63. doi: 10.1093/ckj/sfu034. Epub 2014 Apr 15. PMID 25852886
- [Background] Cook WL, Tomlinson G, Donaldson M, Markowitz SN, Naglie G, Sobolev B, Jassal SV. Falls and fall-related injuries in older dialysis patients. Clin J Am Soc Nephrol. 2006 Nov;1(6):1197-204. doi: 10.2215/CJN.01650506. Epub 2006 Aug 30. PMID 17699348
- [Background] Couch ME, Dittus K, Toth MJ, Willis MS, Guttridge DC, George JR, Barnes CA, Gourin CG, Der-Torossian H. Cancer cachexia update in head and neck cancer: Definitions and diagnostic features. Head Neck. 2015 Apr;37(4):594-604. doi: 10.1002/hed.23599. Epub 2014 Mar 25. PMID 24415363
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334